CLINICAL TRIAL: NCT05967169
Title: Early Feasibility Study of Bioabsorbable Polydioxanone Implant and Delivery Device for Correction of Cartilaginous Septal Deviation
Brief Title: EFS of Bioabsorbable Implant for NSD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spirair, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT-001
Record Dates: First submitted 2023-07-13; First posted 2023-08-01 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Nasal Septal Deviation

STUDY DESIGN:
Intervention Model Description: Multi-cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Cohort 1 (Experimental): Index Procedure in OR, placement of one implant
  Interventions: Device: Nasal Septal Strap implantation
- Cohort 2 (Experimental): Index Procedure in office or OR, placement of one implant
  Interventions: Device: Nasal Septal Strap implantation
- Cohort 3 (Experimental): Index Procedure in OR, placement of up to two implant
  Interventions: Device: Nasal Septal Strap implantation

INTERVENTIONS:
Device: Nasal Septal Strap implantation — Correction of NSD with Nasal Septal Strap implant

SUMMARY:
Early feasibility study of bioabsorbable implant and delivery device for correction of septal deviation

DETAILED DESCRIPTION:
To obtain safety, device performance, patient tolerability and effectiveness outcome data in participants with cartilaginous septal deviations undergoing placement of the Spirair Implant with the Spirair delivery device.

ELIGIBILITY:
Inclusion Criteria:

* Non-calcified, mobile cartilaginous septal deviation.
* ≥21 years of age.
* Willing and able to provide informed consent and comply with the study protocol.
* Seeking treatment for nasal airway obstruction (NAO) due to septal deviation and is willing to undergo a nasal implant procedure.
* Type I, II, or III septal deviation as defined by 7-Degree Mladina classification scheme
* NOSE score ≥30 at Screening Visit.
* Appropriate nasal anatomy to receive the implant(s).

Exclusion Criteria:

* Type IV, V, VI or VII septal deviation as defined by 7-Degree Mladina classification scheme (See Table 2) or other non-cartilaginous septum anatomical pathology identified on CT scan suspected by Investigator to be the primary contributor to NAO.
* Having a concurrent ENT procedure, other than turbinate reduction.
* Previous septoplasty or rhinoplasty.
* Has had turbinate reduction or other nasal surgeries within the past six (6) months.
* Plans to have any surgical or non-surgical treatment of their nasal septum, other than the index procedure, within six (6) months of the procedure.
* Permanent implant or dilator in the nasal area.
* Concomitant autoimmune, inflammatory, or infectious skin conditions, unhealed wounds, septal perforation, or mucosal irregularities in the treatment area.
* Currently has active nasal vestibulitis or folliculitis.
* History of nasal vasculitis.
* Current or chronic systemic steroid and/or recreational intra-nasal drug user.
* Has had a cancerous or pre-cancerous lesion and/or has had radiation exposure in the treatment area or active chemotherapy.
* Polyps or pathology, other than turbinate hypertrophy, that may be primary contributor to airway obstruction, in the opinion of the investigator.
* History of a significant bleeding disorder(s) and/or current prescription blood thinner medication that would prevent healing of the treatment area post procedure.
* Known or suspected allergy to polydioxanone or other absorbable materials.
* Significant systemic disease such as poorly controlled diabetes or connective tissue disease which, in the investigator's opinion, could pre-dispose the participant to poor wound healing.
* Current tobacco or tobacco-related product use or history within the past 10 years of heavy smoking (on average, more than half a pack of cigarettes per day).
* Female participants of childbearing potential who are known or suspected to be pregnant and/or lactating.
* Any physical condition that, in the Investigator's opinion, would prevent adequate study participation or increase risk.
* Additionally, for OR cases (Cohorts 1 or 3) any individual who meets the following criteria will be ineligible for enrollment as an OR case

  * Is not a candidate for procedures conducted under general anesthesia.
* Additionally, for in-office cases (Cohort 2) any individual who meets the following criteria will be ineligible for enrollment as an in-office case:

  * s not a candidate for procedures conducted under local anesthesia alone.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2025-12-08 (Estimated); Study Completion 2025-12-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with successful implantation as measured through physician's assessment and patient reported outcomes | 24 months
  Feasibility of implantation and durability of Implant through the healing process

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Breathe Clear Institute, Torrance, California
  - Specialty Physicians, Bethlehem, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Davis SE, Davis GE. The Safety and Efficacy of a Bioabsorbable Implant for Correction of Cartilaginous Septal Deviation. Ear Nose Throat J. 2025 Jun 4:1455613251346589. doi: 10.1177/01455613251346589. Online ahead of print. PMID 40468718